CLINICAL TRIAL: NCT06597851
Title: Insulin Resistance and Coronary Microvascular Dysfunction in Patients with Myocardial Ischemia and Non-obstructive Coronary Artery Disease
Acronym: IRIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Roberto Scarsini, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRIN (225CET)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Coronary Microvascular Dysfunction; Coronary Microvascular Disease; Insulin Resistance
Keywords: Coronary Microvascular Dysfunction; Coronary Microvascular Disease; Insulin Resistance; INOCA; ANOCA; CMD; hyperinsulinemic-euglycemic clamp test
MeSH Terms: conditions — Microvascular Angina; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Prospective, experimental, single-arm, explorative study. The study aims to perform a functional study of the coronary microcirculation with pressure guides, in patients with angina and non obstructive coronary artery disease. Also a tranthoracic echocardiography will be performed. Following this, the patient will undergo hyperinsulinemic-euglycemic clamp test to evaluate insulin resistance and the metabolic risk. The primary endpoint is to assess the correlation between the index of microcirculatory resistance and the M-value evaluated with clamp test as a measure of insulin resistance. Follow up will continue up to 1 year from enrollment through telephone contacts, outpatient visits and review of clinical data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-diabetic patients with ANOCA (Experimental): * Thermodilution based assessment of coronary microcirculation with the derivation of CFR and IMR
  * Hyperinsulinemic euglycemic clamp for insulin resistance assessment
  Interventions: Diagnostic Test: Thermodilution based assessment of coronary microcirculation; Diagnostic Test: Hyperinsulinemic-euglycemic Clamp test

INTERVENTIONS:
Diagnostic Test: Thermodilution based assessment of coronary microcirculation — Coronary microvascular assessment with the derivation of CFR, IMR and MRR will be performed using a standard pressure/thermodilution guidewire.
Diagnostic Test: Hyperinsulinemic-euglycemic Clamp test — Infusion of insulin and glucose adjusting rate of glucose infusion to maintaine plasma glucose around 90 mg/dL by monitoring plasma glucose levels every 5-10 minutes

SUMMARY:
The goal of this prospective study is to assess the correlation between coronary microvascular disfunction and insulin resistance in patients with INOCA.

Patients with ANOCA and without diabetes will undergo invasive coronary microvascular assessment through coronary angiography and insulin resistance assessment through hyperinsulinemic-euglycemic clamp test.

Patients enrolled in the study will be followed for a period of 2 years to monitor their clinical status.

DETAILED DESCRIPTION:
This is a prospective, experimental, single-center, explorative study designed to assess the correlation between coronary microvascular disfunction and insulin resistance in patients with INOCA.

Patients identified as eligible for the protocol will be asked for written informed consent to participate in the study.

Participants will undergo multimodality diagnostic tests as per standard clinical practice and international recommendations:

1. Fasting glucose, fasting insulin, HOMA index, glycated haemoglobin and oral glucose tolerance test (OGTT) will be assessed to rule out diabetes.
2. Transthoracic echocardiography will be performed to evaluate cardiac function and cardiac remodeling.
3. Coronary angiography will be performed to rule out obstructive CAD defined as angiographic stenosis ≥ 70% of one or more main epicardial coronary arteries (defined as vessels with diameter >2.0 mm) and/or fractional flow reserve (FFR) ≤ 0,80 as indicated by the latest European Guidelines.
4. In case of angiographic evidence of unobstructive CAD, participants will undergo coronary microvascular function assessment using standard coronary pressure guidewire as indicated by the latest European Guidelines according to the recently described Fullphysiology method. If clinically indicated, in case of suspected epicardial or microvascular spasm, endothelial-dependent vasomotor function will be evaluated using a standard vasoreactivity test based on incremental doses of acetylcoline infusion as indicated by the latest European Guidelines.
5. Patients will undergo hyperinsulinemic-euglycemic clamp test at Diabetology Unit of AOUI Verona to evaluate insulin resistance and the metabolic risk. In patients with no clinical concerns, adequate pharmacological washout from betablockers, ace inhibitors, sartans and/or calcium antagonists will be considered before performing the clamp test.
6. Patients will undergo clinical follow up at 6 and 12 months via outpatient clinic or telephone contacts. Fasting glucose, fasting insulin, HOMA index and glycated haemoglobin will be re-assessed at 12 months.
7. Transthoracic echocardiography will be repeated at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years.
* Cardiac chest pain with evidence of myocardial ischemia at noninvasive myocardial stress imaging and clinical indication to diagnostic coronary angiography
* Willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Obstructive CAD (defined as more than 70% luminal stenosis and/or FFR ≤0.80 in 1 or more epicardial vessels).
* History of previous myocardial infarction, percutaneous revascularization or coronary-aortic bypass graft (CABG) surgery.
* Diagnosis of type II diabetes.
* BMI ≥ 35 kg/m2.
* Stage IV and V of chronic kidney disease (eGFR ≤ 30 ml/min, estimated through CKD - EPI Creatinine Equation).
* Allergy or other contraindication to iodinated contrast and/or gadolinium and/or adenosine.
* Chronic resting O2 saturation ≤ 85%.
* Pregnancy or suspected pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between coronary microvascular dysfunction and insulin resistance | At baseline
  Correlation between the index of microcirculatory resistance (IMR) and the M-value evaluated with the hyperinsulinemic-euglycemic clamp test as a measure of insulin resistance

SECONDARY OUTCOMES:
Correlation in vasomotor function in patients with and without IR | At baseline
  Difference in vasomotor dysfunction at vasoreactivity test with acetylcholine in patients with and without IR
Adverse clinical events | 12 months
  Composite of cardiovascular death, new hospitalization for HF and/or ACS during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Scarsini MD PhD, Principal Investigator — Azienda Ospedaliera Universitaria di Verona
Locations (1):
- Azienda Ospedaliera Universitaria di Verona, Verona, VR, Italy

IPD SHARING:
Plan to Share IPD: Undecided